CLINICAL TRIAL: NCT02069743
Title: Pain Management in Cancer Patients Using a Mobile Application
Acronym: ePAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McKesson Foundation (Other)
Responsible Party: Principal Investigator, Mihir M. Kamdar,M.D., Attending Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-080
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Cancer
Keywords: cancer pain
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will use the study's mobile application during the 8-week study.
  Interventions: Other: ePAL Mobile Application
- Control (No Intervention): The control group will not use the study's mobile application during the study.

INTERVENTIONS:
Other: ePAL Mobile Application — A mobile application designed to help cancer patients better self-manage cancer pain.
  Other Names: ePAL
  Arms: Intervention

SUMMARY:
The investigators have developed a mobile application (for use on smart phones) to help cancer patients better manage cancer pain. This study is a randomized controlled trial to evaluate the effect of this mobile-based intervention. The investigators' hypothesis is that subjects randomized to the intervention group will have a reduction in pain and pain-related hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, 18 years and above suffering from solid-organ cancer.
* Diagnosed with moderate or severe cancer pain (i.e. pain intensity score of at least 4/10 on numeric rating scale (NRS)) at the Massachusetts General Hospital (MGH) Palliative Care Center, as determined by the patient's care provider at the MGH Palliative Care Center. Subjects do not need to experience a specific nature of pain for eligibility.
* Patients must be ambulatory and not currently admitted to the hospital at time of enrollment.
* Must have a smart phone and be willing to download the study application (Phase II only)
* Must be able to read and speak English.

Exclusion Criteria:

* Life expectancy less than 2-months as determined by the palliative care provider
* Significant medical or psychiatric co-morbidities (other than depression or anxiety) or cognitive impediments that would prevent participant from being able to utilize the program
* Known history of substance abuse
* Patients currently on investigational therapies or other study protocols that may have an impact on pain intensity or quality of life which are main outcomes of this intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Pain symptoms using the Brief Pain Inventory | up to 8 weeks
  The primary aim is to assess the effect of a tailored, multi-dimensional mobile-based intervention on the intensity of cancer pain in cancer patients with moderate to severe pain.

SECONDARY OUTCOMES:
Pain related hospitalization from the Electronic Health Record | up to 8 weeks
  * In-patient and out-patient hospital visits
  * Urgent non-scheduled clinic visits for pain crisis
Patient-related barriers to pain management using the Barriers Questionnaire-II | up to 8 weeks
  compared patient-related barriers to pain management using the Barriers Questionnaire-II (BQ-II)
Engagement as tracked by the app | up to 8 weeks
  Pattern of patient engagement with the study's mobile application
Anxiety symptoms using the Generalized Anxiety Disorder (GAD-7) | up to 8 weeks
  compare anxiety symptoms between the two group using the Generalized Anxiety Disorder (GAD-7)
Quality of life using the Functional Assessment of Cancer Therapy (FACT-G) | up to 8 weeks
  to compare quality of life between the two groups using the Functional Assessment of Cancer Therapy -General (FACT-G)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - The Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Agboola S, Kamdar M, Flanagan C, Searl M, Traeger L, Kvedar J, Jethwani K. Pain management in cancer patients using a mobile app: study design of a randomized controlled trial. JMIR Res Protoc. 2014 Dec 12;3(4):e76. doi: 10.2196/resprot.3957. PMID 25500281